CLINICAL TRIAL: NCT01467804
Title: Randomized Double Blinding Controlled Study on" Jia Wei Xiao Yao Jiaonang" Treating Mild to Moderate Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Su Rui (Other)
Responsible Party: Sponsor-Investigator, Su Rui, assistant researcher, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: y00741015-zjx
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2010-01

CONDITIONS: Depressive Disorder
Keywords: efficacy,; safety,; JWXYJN
MeSH Terms: conditions — Depressive Disorder | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese medicine (Experimental): There are 90 patients with mild to moderate depress in JWXY group, who take the JWXY capsule, and placebo of Sertraline, for 2 months
  Interventions: Drug: JWXYJN plus placebo of Sertraline
- westen medicine (Active Comparator): There are 90 patients with mild to moderate depress in westen medicine group, who take Sertraline, and placebo of the JWXY capsule, for 2 months
  Interventions: Drug: Sertraline plus placebo of JWXYJN

INTERVENTIONS:
Drug: Sertraline plus placebo of JWXYJN — oral sertraline (start with 50 mg/day for one week then continue with 100 mg/day plus placebo of JWXYJN
  Arms: westen medicine
Drug: JWXYJN plus placebo of Sertraline — JWXYJN 3.6g/d plus placebo of sertraline
  Arms: Chinese medicine

SUMMARY:
This is a randomized, double-blind multi centric clinic study. Both of therapist and patient are blind. There are 180 patients from 3 hospitals included, who meet DSM-IV criteria for major depressive disorder, the score of HAMD-item>20，<35；and meet the criteria for TCM syndrome of "Liver Qi stagnation and Transformation of Stagnant Qi into Fire". Patients are randomized to JWXY and sertraline treatment groups, receiving oral sertraline (start with 50 mg/day for one week then continue with 50 mg/day) plus placebo of JWXYJN; or oral JWXYJN plus placebo of sertraline daily for 2 months. The symptoms of depression and anxiety are measured with HAMD and HAMA tests at baseline and at 2，4，8 weeks; and LFT, BUN, Cr are assessed at baseline and end of program. Then data will be analyzed with SPSS software to determine the efficacy and safety of JWXYJN comparing to sertraline in the treatment of mild to moderate major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* A diagnosis of MDD, single episode or recurrent, according to DSM-IV
* Meets DSM-IV criteria for Major Depressive Disorder.
* factor score from the 24-item Hamilton Depression Rating Scale (HAM-D) >20,<35
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Patients with a current (or within 6 months prior to the Screening Visit) Axis I disorder of Post Traumatic Stress Disorder, Eating Disorder, Obsessive Compulsive Disorder.
* Patients with a history of schizophrenia, schizoaffective disorder or bipolar I or II disorder (with a history of hypomanic or manic episodes).
* Patients who meet DSM-IV criteria for substance abuse (alcohol or drugs) within 3 months prior to Screening Visit or substance dependence within 6 months prior to the Screening Visit.
* Patients who meet criteria for any of the following DSM-IV MDD Specifiers: [a] With Catatonic Features; [b] With Postpartum Onset; [c] With Seasonal Pattern [d] with Psychotic Features.
* Patients who are receiving formal psychotherapy or have had psychotherapy within the 12 weeks prior to the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
HAMD scale | 12 weeks
  HAMD scale to access the depression level

CONTACTS AND LOCATIONS:
Locations (1):
- China Academy of Chinese Medicine Science, Beijing, Beijing Municipality, China